CLINICAL TRIAL: NCT05606328
Title: Improving Delirium Screening and Detection for Older Adults Presenting to the Emergency Department (ED): A Novel ED Delirium Screening and Detection Program
Brief Title: Implementation Outcome Assessments of the Emergency Department Delirium Screening and Detection Program
Acronym: ED-DDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0681; R21AG075230 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Delirium
Keywords: Delirium Screening; Delirium Detection; Emergency Department; Older Adults
MeSH Terms: conditions — Delirium; Emergencies

STUDY DESIGN:
Intervention Model Description: This study is a pilot stepped wedge cluster randomized trial (SW-CRT) of three diverse emergency department (EDs) randomized to receive the intervention at 3-month intervals over a 15-month period. Time of crossover from the control to intervention period will be unidirectional, and each crossover sequence will allow for a 3-month implementation period where data will not be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation Period (Experimental): ED leadership at each site will identify 5-10 delirium champions (nurse educators and managers, bedside nurses) based on their interest in delirium and commitment to program participation, including training of nurses by champions. The implementation period will take place over a period of 3 months. No data analysis will take place during the implementation period.
  Interventions: Behavioral: Emergency Department Delirium Screening and Detection Program (ED-DDP)
- Intervention Period (No Intervention): The intervention period will take place 3-9 months after implementation of the ED-DDP program over a 15 month period, depending on when a site is randomized to receive the ED-DDP intervention.

INTERVENTIONS:
Behavioral: Emergency Department Delirium Screening and Detection Program (ED-DDP) — Champions will participate in a 1-day workshop, consisting of patient testimonials, small group discussions, delirium and screening tool use (didactics), and role-playing. Following the workshop, champions will receive 3 tele-training sessions; 2 to provide direct observation/feedback while the champion performs a bedside delirium screen, and 1 to provide direct observation/feedback of the champion providing training to the nurse. Once delirium champions complete training, they will provide bedside delirium training for all ED nurses. No adaptations to the ED-DDP will occur between implementation sites and no data will be collected during implementation phases.
  Arms: Implementation Period

SUMMARY:
Delirium occurs in up to 20% of older adults presenting to the Emergency Department (ED) and is associated with poor outcomes. Failure to identify patients with ED delirium not only prevents initiation of mitigation strategies, but is also a barrier to advancing the field in terms of evaluating management and clinical outcomes. This project studies the potential of an ED Delirium Detection Program (ED-DDP), developed to address the need for consistent and accurate ED delirium detection.

This research will have two objectives:

* Aim 1 will conduct a pilot stepped wedge cluster randomized trial (SW-CRT) of the ED-DDP across 3 diverse EDs to determine preliminary efficacy of the detection training program, and
* Aim 2 will use a mixed methods approach to assess RE-AIM implementation outcomes (Reach, Efficacy, Adoption, Implementation, and Maintenance) of the training program.

Aim 1 will consist of a multicomponent 1-day delirium champion workshop where the training is delivered, real-time direct observation/training of champions via telehealth, practical training of nurses throughout each ED by champions, and patient chart review. In Aim 2, the investigators will assess implementation outcomes using training logs, tele-observation, interviews with champions and nurses, and electronic medical record screening.

The overarching aim of this proposal is to determine the preliminary efficacy of the training program for improving ED delirium screening, detection, and management in older adults, while also evaluating implementation outcomes of the program for champions/nurses. The investigators will use findings from this study to inform a full-scale SW-CRT to evaluate the impact of the program on patient outcomes at Northwell Health. The long-term goal of this study is to implement and disseminate a comprehensive ED-DDP that will improve screening, detection, and management of ED delirium in older adults.

DETAILED DESCRIPTION:
Grounded in the RE-AIM framework, investigators will use mixed methods to conduct implementation outcome assessments of the ED-DDP for champions and nurses. A multimodal approach, using training logs, tele-observations, and EHR data, will assess quantitative outcomes during implementation/intervention periods: Reach (training completion), Efficacy (accurate screening tool use), Adoption (screening rates), and Implementation (fidelity/time of program delivery). Investigators will conduct semi-structured interviews (intervention period) to assess and explain: successes and challenges of training completion (Reach) and Adoption of delirium screening; adaptations made to ED DDP delivery (Implementation); and plan for Maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Nurse educators, managers, or bedside nurses self-identified or recommended by emergency department (ED) leadership to volunteer as a program site champion
* Primarily working at a participating ED site
* Commitment to program participation

Exclusion Criteria:

* Unable to meet program requirements, including attending champion workshop, agreement to observation and training via telehealth, and commitment to train department staff
* Does not primarily work in the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Sinvani, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institutes for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospital Site A Nurse Champions: The Emergency Department Delirium Screening and Detection Program (ED-DDP) intervention consisted of enrollment of Nurse Champion participants at participating ED sites. Nurse Champions were identified by site leaders before approaching for enrollment. All Nurse Champions received a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during their site's Implementation Period. Participant flow is reported during the Implementation Period only, as this is when all program components started and completed for each enrolled participant. The Emergency Department in Hospital Site A received the Implementation Period during months 4-6.
- Hospital Site B Nurse Champions: The Emergency Department Delirium Screening and Detection Program (ED-DDP) intervention consisted of enrollment of Nurse Champion participants at participating ED sites. Nurse Champions were identified by site leaders before approaching for enrollment. All Nurse Champions received a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during their site's Implementation Period. Participant flow is reported during the Implementation Period only, as this is when all program components started and completed for each enrolled participant. The Emergency Department in Hospital Site B received the Implementation Period during months 7-9.
- Hospital Site C Nurse Champions: The Emergency Department Delirium Screening and Detection Program (ED-DDP) intervention consisted of enrollment of Nurse Champion participants at participating ED sites. Nurse Champions were identified by site leaders before approaching for enrollment. All Nurse Champions received a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during their site's Implementation Period. Participant flow is reported during the Implementation Period only, as this is when all program components started and completed for each enrolled participant. The Emergency Department in Hospital Site C received the Implementation Period during months 10-12.
Period: Months 1-3
Arm/Group | Hospital Site A Nurse Champions | Hospital Site B Nurse Champions | Hospital Site C Nurse Champions
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Months 4-6
Arm/Group | Hospital Site A Nurse Champions | Hospital Site B Nurse Champions | Hospital Site C Nurse Champions
Started (Of note, Nurse Champions started and completed the Delirium Detection Program during 1 period. No new Nurse Champions started the program in subsequent periods. Cumulative numbers are reported. Hospital A: Period 1: control; Period 2: implementation; Periods 3-5: intervention Hospital B: Periods 1-2: control; Period 3: implementation; Periods 4-5: intervention Hospital C: Periods 1-3: control; Period 4: implementation; Period 5: intervention) | 6 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 1 | 0 | 0
Period: Months 7-9
Arm/Group | Hospital Site A Nurse Champions | Hospital Site B Nurse Champions | Hospital Site C Nurse Champions
Started | 6 | 6 | 0
Completed | 5 | 6 | 0
Not Completed | 1 | 0 | 0
Period: Months 10-12
Arm/Group | Hospital Site A Nurse Champions | Hospital Site B Nurse Champions | Hospital Site C Nurse Champions
Started | 6 | 6 | 6
Completed | 5 | 6 | 6
Not Completed | 1 | 0 | 0
Period: Months 13-15
Arm/Group | Hospital Site A Nurse Champions | Hospital Site B Nurse Champions | Hospital Site C Nurse Champions
Started | 6 | 6 | 6
Completed | 5 | 6 | 6
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nurse champions enrolled in the ED-DDP program.
Groups:
- Hospital Site A: The Emergency Department in Hospital Site A received the following study sequence: 3 month Control Period, then a 3 month Implementation Period, then a 9 month Intervention Period. The Emergency Department Delirium Screening and Detection Program (ED-DDP) was delivered during Implementation Period only and consisted of identification and enrollment of Nurse Champion participants to receive a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during the Implementation Period. Pre and post program data was collected during the Control Period and Intervention Period, respectively.
- Hospital Site B: The Emergency Department in Hospital Site B received the following study sequence: 6 month Control Period, then a 3 month Implementation Period, then a 6 month Intervention Period. The Emergency Department Delirium Screening and Detection Program (ED-DDP) was delivered during Implementation Period only and consisted of identification and enrollment of Nurse Champion participants to receive a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during the Implementation Period. Pre and post program data was collected during the Control Period and Intervention Period, respectively.
- Hospital Site C: The Emergency Department in Hospital Site C received the following study sequence: 9 month Control Period, then a 3 month Implementation Period, then a 3 month Intervention Period. The Emergency Department Delirium Screening and Detection Program (ED-DDP) was delivered during Implementation Period only and consisted of identification and enrollment of Nurse Champion participants to receive a 1-day workshop and 3 tele-training sessions. Once Nurse Champions completed trainings, they provided baseline delirium training to all nurses at their site Emergency Department during the Implementation Period. Pre and post program data was collected during the Control Period and Intervention Period, respectively.
- Total: Total of all reporting groups
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 14
  Male | 0 | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 1 | 6 | 3 | 10
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 2
Years of Practice [Number; unit: Years] — Number of years of experience as a nurse.
  Years
    1-5 Years | 0 | 1 | 3 | 4
    6-10 Years | 1 | 5 | 1 | 7
    11-15 Years | 1 | 0 | 1 | 2
    Over 15 Years | 4 | 0 | 1 | 5
Education [Count of Participants; unit: Participants] — Highest level of educational degree obtained.
  Participants
    BS/BA | 2 | 5 | 4 | 11
    MS/MA | 2 | 1 | 1 | 4
    PhD/EdD/SciD | 1 | 0 | 0 | 1
    Practice doctorate (MD, DNP, etc.) | 0 | 0 | 1 | 1
    Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Accurate Delirium Screening by Emergency Department (ED) Nurses (RE-AIM: Efficacy)
Description: Tele-observations will be used to asses screening accuracy, defined as the proportion of nurses who score at least 80% accuracy on the brief confusion assessment method (bCAM) use using a validated Spot Check Form. The investigators will observe a random sample of nurses (N=30, 10 at each ED site) performing a delirium screen in real-time. A successful outcome will be considered if computed proportion of nurses accurately using the bCAM tool is 80% or higher.
Time Frame: Intervention period (3-9 months post program implementation)
Population: Site nurses were not considered enrolled in the study but were assessed for this measure.
Measure: Count of Units; unit: Site nurses who received Spot Check Form
Units Other Than Participants: Site nurses who received Spot Check Form
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 5 | 6 | 6
Number analyzed (Site nurses who received Spot Check Form) | 10 | 10 | 10
Site nurses who received Spot Check Form | 4 | 1 | 8

2. Secondary Outcome: Proportion of Delirium Champions Who Complete Training (RE:AIM: Reach)
Description: Champion training logs will be used to determine the proportion of champions who complete training (1-day workshop and 3 tele-training sessions) at each emergency department site. A successful outcome will be considered if computed proportion is 80% or higher.
Time Frame: Implementation period (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 6 | 6 | 6
Participants | 5 | 6 | 6

3. Secondary Outcome: Proportion of Emergency Department Nurses Who Complete Training (RE-AIM: Reach)
Description: Emergency department nurse training logs will be used to determine the proportion of nurses who complete at least 1 training session with a delirium champion at each ED site. A successful outcome will be considered if computed proportion is 80% or higher.
Time Frame: Implementation period (3 months)
Population: Site nurses were not considered enrolled in the study but were assessed for this measure.
Measure: Count of Units; unit: Total number of nurses at site
Units Other Than Participants: Total number of nurses at site
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 5 | 6 | 6
Number analyzed (Total number of nurses at site) | 46 | 73 | 100
Total number of nurses at site | 46 | 66 | 83

4. Secondary Outcome: Proportion of Nurses Who Screen Eligible Patients (REAIM: Adoption)
Description: Electronic health record (EHR) data will be used to determine the proportion of nurses who document delirium screening in at least 80% of eligible patients. A successful outcome will be considered if computed proportion is 80% or higher. Data is reported as the number of patient records reviewed during the intervention period that contained a delirium screening by a emergency department nurse.
Time Frame: Intervention period (3-9 months post implementation)
Measure: Count of Units; unit: Electronic health records reviewed
Units Other Than Participants: Electronic health records reviewed
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 5 | 6 | 6
Number analyzed (Electronic health records reviewed) | 747 | 497 | 248
Electronic health records reviewed | 450 | 9 | 39

5. Secondary Outcome: Proportion of Training Program Components That Adhered to ED-DDP Protocol (REAIM: Implementation/Fidelity)
Description: Training logs of delirium champions and ED nurses will be used to determine the proportion of training components (workshop, tele-training sessions, and bedside training of nurses by champions) that adhered to ED-DDP protocol. A successful outcome will be considered if computed proportion is 80% or higher.
Time Frame: Implementation period (3 months)
Measure: Count of Units; unit: Training Components
Units Other Than Participants: Training Components
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 6 | 6 | 6
Number analyzed (Training Components) | 6 | 6 | 6
Training Components | 5 | 6 | 6

6. Secondary Outcome: Time Required to Train Delirium Champions and Nurses (REAIM: Implementation/Time)
Description: Data is reported as total number of days necessary to train 80% of nurses in the ED site. Training logs of delirium champions and ED nurses will be used to determine the time required to complete champion and ED nurse training. A successful outcome will be considered if 80% of delirium champion and ED nurses complete training within the implementation period (fewer than 90 days).
Time Frame: Implementation period (3 months)
Population: Site nurses were not considered enrolled in the study but were assessed for this measure.
Measure: Number; unit: Days
Units Other Than Participants: Total number of nurses at site
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
Number analyzed (Participants) | 5 | 6 | 6
Number analyzed (Total number of nurses at site) | 46 | 73 | 100
Days | 72 | 72 | 49

ADVERSE EVENTS:
Time Frame: During the 3-Month Implementation Period
Arm/Group | Hospital Site A | Hospital Site B | Hospital Site C
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05606328/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05606328/ICF_001.pdf